CLINICAL TRIAL: NCT06062524
Title: Guo's False Lumen Embolization : The First in Man Study of WeFlow-EndoSeal Aorta Vascular Plug System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endoseal V1.0
Record Dates: First submitted 2023-09-15; First posted 2023-10-02 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-09

CONDITIONS: Aortic Dissection Aneurysm
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-EndoSeal Aorta Vascular Plug System (Experimental): WeFlow-EndoSeal Aorta Vascular Plug System
  Interventions: Device: Aorta Vascular Plug System

INTERVENTIONS:
Device: Aorta Vascular Plug System — The Aorta Vascular Plug System for false lumen is composed of a vascular plug system and an adjustable bend conveyor. The plug system is composed of a patch and a conveying steel cable. The plug is pre-installed on the conveying steel cable.

SUMMARY:
A prospective, single-center, first in man study to evaluate the safety and efficacy of WeFlow-EndoSeal Aorta Vascular Plug System manufactured by Hangzhou Endonom Medtech Co., Ltd. for the dissecting aneurysm of descending thoracic aorta after aortic dissection repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years old, no gender limitation;
* The patient was diagnosed with a dissecting aneurysm of the descending thoracic aorta after the repair of the main artery dissection, and the treatment indications were one of the following:

  1. Aortic dissection aneurysm diameter ≥ 5.5cm
  2. The diameter of descending thoracic aorta dissection increased rapidly ≥5 mm/ year
  3. Symptoms associated with dissection progression, such as chest and back pain
* The diameter of false lumen approximately 1 cm superiorly to the celiac trunk ≤40 mm
* Appropriate anatomical conditions were assessed by imaging to allow the adjustable bend conveyor to enter the pseudolumen through tears of the iliac artery, subrenal aorta, or renal artery levels.
* Those who can understand the purpose of the trial, voluntarily participate in the study, sign the informed consent form by themselves or their legal representative, and are willing to complete the follow-up according to the protocol requirements.

Exclusion Criteria:

* Aortic rupture;
* Continuous malperfusion of internal artery branches caused by dissection;
* Had previously received false lumen embolization;
* Proximal type I endoleak after aortic repair;
* Abdominal aortic dissection aneurysm diameter > 5 cm
* Infectious aortic disease, arteritis, Marfan syndrome (or other connective tissue diseases);
* Acute systemic infection;
* History of myocardial infarction, TIA or cerebral infarction within the past 3 months;
* Cardiac function Grade IV (NYHA rating) or LVEF < 30%;
* Hematological abnormalities: leukopenia (WBC < 3×10^9/L), anemia (Hb < 90 g/L); Coagulation dysfunction, thrombocytopenia (PLT count < 50×10^9/L);
* Renal insufficiency: serum creatinine > 150 umol/L (or 3.0 mg/dL) and/or advanced kidney disease requiring renal dialysis, as determined by the investigator after thorough analysis;
* Severe liver insufficiency: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds the normal upper limit by 5 times; Serum total bilirubin (STB) exceeded the normal upper limit by 2 times;
* Allergic to contrast agents, anesthetics, plugs, and delivery materials;
* Pregnant, breastfeeding or cannot contraception during the trial period;
* Participated in clinical trials of other drugs or devices during the same period;
* Life expectancy is less than 12 months (such as advanced malignant tumors);
* Investigator judged that not suitable for interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
No major adverse events within 30 days after operation. | 30 days after operation
  Major adverse events within 30 days after operation refer to all-cause death, myocardial infarction, ischemic stroke, respiratory failure, renal failure, intestinal necrosis, paraplegia, and amputation within 30 days after operation. Among them, renal failure refers to long-lasting dialysis, kidney transplantation, or other fatal results. Intestinal necrosis is intestinal ischemia that requires bowel resection or other fatal consequences. Severe lower limb ischemia refers to new severe limp or resting pain after surgery.
All-cause mortality | 30 days, 6 months, and 12 months after operation
  All-cause mortality includes cardiac mortality, non-cardiac mortality, and mortality from unknown causes.
Aortic dissection-related mortality, | 30 days, 6 months, and 12 months after operation
  Refers to mortality caused by a ruptured aortic dissection or endovascular interventional treatment.
Serious adverse events. | 30 days, 6 months, and 12 months after operation
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.
False lumen thrombosis of the descending thoracic aorta | 1 month, 6 months, and 12 months after operation
  False lumen thrombosis of the descending thoracic aorta (no thrombosis, partial thrombosis, complete thrombosis) observed by postoperative CTA review.
Aortic dissection progression under control | 1 month, 6 months, and 12 months after operation
  Aortic dissection progression under control is defined as maximum increase in the diameter of false lumen diameter in descending thoracic aorta was ≤ 5 mm when compared with preoperative aortic dissection as of postoperative CTA review.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese PLA Gencral Hosptial, Beijing, Beijing Municipality
  - The People's Hospital of Gaozhou, Gaozhou, Guangdong
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided